CLINICAL TRIAL: NCT07344454
Title: STORK (Supporting the Transition to Parenthood Through Online Sex and Relationship Knowledge) Randomized Controlled Trial
Brief Title: Supporting the Transition to Parenthood Through Online Sex and Relationship Knowledge
Acronym: STORK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Natalie Rosen, Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-7940; 435-2023-0235 (Other Grant/Funding Number: Social Sciences and Humanities Research Council of Canada (SSHRC))
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy; Postpartum
Keywords: Transition to parenthood; sexual well-being; couples; parents

STUDY DESIGN:
Intervention Model Description: The randomized controlled trial will evaluate the efficacy of a novel 6-module online psychoeducational program (STORK) for couples undergoing the transition to parenthood compared to a waitlist control group. Couples in the program (i.e., experimental) group will receive access to the STORK program. Couples in the waitlist control group will complete all questionnaires at the equivalent timepoints as the experimental group and, at the end of the 12-month follow-up, will also receive access to the STORK program for 6 months at no cost.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A free randomization software (www.studyrandomizer.com) will be used for randomization. At each site, allocation will be computer-generated randomly using permuted blocks of size 6 (fixed) to maintain equilibrium between the two conditions (experimental and control). Participants will be instructed not to reveal the condition they are in to the researchers. To that end, participants in the experimental condition will be instructed to contact a separate email address for questions concerning the STORK program that does not go to the main study email. This procedure ensures that the personnel conducting reminder calls for the surveys or conversing with participants via email will not be aware of participant condition and that the PIs will not influence the randomization process. Only the research coordinators (one per site) conducting the randomizations and the STORK facilitators who support couples in the experimental condition will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STORK Program (Experimental): STORK online prevention program
  Interventions: Other: STORK Program
- Waitlist Control (No Intervention): Waitlist control comparison group

INTERVENTIONS:
Other: STORK Program — The STORK program includes a brief orientation module (Module 0, intended to be completed in the same sitting as Module 1) followed by six full-length modules: five weekly modules in pregnancy (Modules 1 to 5) and one module at 3-months postpartum (Module 6). Couples are assigned a trained facilitator (undergraduate research assistant, graduate student, or postdoc) to answer questions or resolve any technical issues.
  Arms: STORK Program

SUMMARY:
Becoming parents exerts powerful and long-lasting effects on couples' well-being and quality of life. The transition to parenthood (TtP; pregnancy to 12-months postpartum) poses significant challenges as couples balance the task of caring for a newborn while maintaining their romantic relationship. One crucial way that couples sustain their connection is through their sexuality. Most new parents experience significant disruptions to their sexual well-being (i.e., sexual satisfaction, desire, distress), with sexual concerns such as reduced sexual frequency and lack of time and energy for sex being nearly ubiquitous. Simultaneously, most new parents lack easily accessible, reliable information on the common sexual changes associated with the TtP and there is a lack of evidence-based research aimed at helping couples navigate changes to their sexual well-being across this life transition. The investigators have identified risk (e.g., stress) and protective (e.g., intimacy) factors for couples' sexual well-being across the TtP that can be targeted in a prevention program, though no such programs exist.

The goal of this two-centre randomized controlled trial is to evaluate the efficacy of STORK (Supporting the Transition to Parenthood through Online Sex and Relationship Knowledge), a novel couple-based online program to support new parents' sexual well-being. This program comprises psychoeducation about common sexual changes as well as skills that couples can develop together to manage these changes and constitutes the first evidence-based program for new parent couples' sexual well-being. The investigators expect that, compared to a waitlist control group, couples who complete STORK will have better sexual, relational, and psychological adjustment across the transition to parenthood (from 13 to 27-weeks gestation to 12-months postpartum). Given that up to 78% of new parents report receiving little-to-no information about what to expect regarding changes to their postpartum sexual relationship, this study addresses the need for accessible, couple-based supports for this commonly challenging transition. By strengthening couples' sexual relationships, the results of this research have the potential to promote the quality of new parents' relationships, strengthening the overall well-being of their families during this critical life stage.

DETAILED DESCRIPTION:
Becoming parents exerts powerful and long-lasting effects on couples' well-being and quality of life. The transition to parenthood (TtP; pregnancy to 12-months postpartum) poses significant challenges as couples balance the task of caring for a newborn while maintaining their romantic relationship. One crucial way that couples sustain their connection is through their sexuality. Sexual satisfaction is one of the top five predictors of relationship quality and is linked to lower perinatal anxiety, depression, and stress-all of which affect children's socioemotional development. Most new parents experience significant disruptions to their sexual well-being (i.e., sexual satisfaction, desire, distress), with sexual concerns such as reduced sexual frequency and lack of time and energy for sex being nearly ubiquitous. Simultaneously, most new parents lack easily accessible, reliable information on the common sexual changes associated with the TtP. Indeed, up to 78% of new parents report receiving little-to-no information about what to expect regarding changes to their postpartum sexual relationship. However, this information is fundamental to establish realistic expectations and to successfully manage the sexual changes likely to occur. There is a lack of evidence-based research aimed at helping couples navigate changes to their sexual well-being across this life transition. Studies that do exist are small, atheoretical, lack postpartum follow-up and typically focus on new mothers, neglecting partners' experiences as well as the interdependency of couples' sexuality. The investigators have identified risk (e.g., stress) and protective (e.g., intimacy) factors for couples' sexual well-being across the TtP that can be targeted in a prevention program, though no such programs exist.

The investigators have subsequently developed STORK (Supporting the Transition to Parenthood through Online Sex and Relationship Knowledge), a couple-based online program to support new parents' sexual well-being. STORK is rooted in scientific evidence drawn from our prior research identifying relevant protective and risk factors that are associated with changes in sexual well-being during the TtP. The program comprises psychoeducation about common sexual changes as well as skills that couples can develop together to manage these changes and constitutes the first evidence-based program for new parent couples' sexual well-being. The current study builds on a pilot study that found the STORK program was feasible and useful and supported the sexual well-being of new-parent couples from mid-pregnancy to 3-months postpartum.

The primary aim is to test the prediction that the STORK program will show efficacy in supporting the sexual adjustment of couples in the TtP, such that couples in the program group will report greater sexual satisfaction and desire and lower sexual distress at follow-up (4-months postpartum) and across the postpartum period (4, 8, and 12 months) relative to the control group. As the secondary aim, it is also predicted that couples in the program group will report better relational (i.e., greater relationship satisfaction and less relationship and sexual conflict) and psychological well-being (i.e., less symptoms of depression, anxiety) at follow-up (4-months postpartum) and across the postpartum period (4, 8, and 12 months) relative to the control group.

The investigators will (1) recruit an inclusive sample of 268 first-time expectant couples in their second trimester (13-27 weeks) of pregnancy; (2) randomize couples to either the STORK program or a waitlist control group; (3) have couples complete standardized, self-report measures at baseline (pre-program), 32-weeks gestation, 4-, 8-, and 12-months postpartum; (4) test the efficacy of STORK compared to the control group. Procedures will take place at Dalhousie University and the University of British Columbia.

This clinical trial addresses an important need for empirically validated, accessible, couple-based supports for the transition to parenthood-a time where couples commonly experience new sexual and relationship challenges. By strengthening couples' sexual relationships, the current research program has the potential to promote the quality of new parents' relationships, strengthening the overall well-being of their families during this critical life stage.

ELIGIBILITY:
Inclusion Criteria:

* married or cohabitating romantic relationship of at least 12 months
* one member of the couple must be currently pregnant (13-27 weeks gestation) with their first baby together (If the couple has a history of miscarriage or stillbirth, previously gave a baby up for adoption, or have other children who do not live with them, they are still eligible to participate.)
* low-risk pregnancy
* live in Canada, the United States, Australia, New Zealand, the Republic of Ireland, or the United Kingdom
* able to read and understand English
* have access to a personal e-mail account

Exclusion Criteria:

* severe relational distress or conflict as determined by baseline measures
* one or both partners of a couple do not complete the baseline survey - this includes cases where one or both partners do not pass at least 3/5 attention checks in the baseline survey
* instructed to avoid sexual activity from a healthcare professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Sexual Satisfaction | Baseline, 32-weeks gestation, and 4-, 8-, and 12-month follow-ups
  The Global Measure of Sexual Satisfaction Scale consists of five items assessing a subjective evaluation of the sexual relationship: good vs. bad, pleasant vs. unpleasant, positive vs. negative, satisfying vs. unsatisfying, and valuable vs. worthless (Lawrance & Byers, 1995). Ratings are summed where possible scores range from 5 to 35, with higher scores indicating greater sexual satisfaction. This measure has demonstrated excellent psychometrics in previous studies (e.g., Paquette et al., 2025).
Sexual Distress | Baseline, 32-weeks gestation, and 4-, 8-, and 12-month follow-ups
  Sexual distress will be assessed with the 3-item Sexual Distress Scale-3 (Derogatis, 2008; Lin et al., 2024). Using a 5-point Likert scale, participants rate how frequently (e.g., 0 = never, to 4 = always) they experience a sexuality related problem. Ratings are summed such that possible scores range from 0 to 12, with higher scores indicating greater sexual distress. This measure has demonstrated good psychometrics in differentiated individuals who did and did not experience sexual problems (Lin et al., 2024).
Sexual Desire | Baseline, 32-weeks gestation, and 4-, 8-, and 12-month follow-ups
  Sexual desire will be measured using 7-items of partner-focused sexual desire from the Sexual Desire Inventory (Moyano et al., 2017). Participants rate their interest in sexual activity using a Likert-type response scale from 0 (e.g., not at all) to 7 or 8 (e.g., a lot). Ratings are summed (range = 0 to 54) such that higher scores indicate greater sexual desire for one's partner. This measure has demonstrated good psychometrics (Moyano et al., 2017).

SECONDARY OUTCOMES:
Depressive Symptoms | Baseline, 32-weeks gestation, and 4-, 8-, and 12-month follow-ups
  The Edinburgh Postnatal Depression Scale (EPDS; Cox, 1987) is a widely used 10-item measure designed to screen for perinatal depression in pregnancy and in parents with infants. The EPDS asks individuals to answer how they have been feeling in the previous 7 days using a response scale from 0 (e.g., Not at all) to 3 (e.g., As much as I ever did), with questions involving common indicators of depression. A total sum score is computed (range = 0 to 30) where higher scores indicate more depressive symptoms. This measure has good psychometric properties (e.g., Kernot et al., 2014) and high sensitivity for detecting postnatal depression (e.g., Eberhard-Gran et al., 2001).
Anxiety Symptoms | Baseline, 32-weeks gestation, and 4-, 8-, and 12-month follow-ups
  Anxiety symptoms will be measured using the 7-item GAD-7 (Spitzer et al., 2006), which assesses symptoms of generalized anxiety. Participants rate the frequency of experiencing anxiety symptoms on a Likert scale from 0 (Not at all) to 3 (Nearly every day). A total sum score is computed (range = 0 to 21) with higher scores indicating greater anxiety symptoms. This measure has good psychometric properties (Spitzer et al., 2006).
Relationship Satisfaction | Baseline, 32-weeks gestation, and 4-, 8-, and 12-month follow-ups
  Relationship satisfaction will be measured with the 4-item version of the Couples Satisfaction Index (CSI) developed by Funk and Rogge (Funk, 2007). Participants rate their general relationship satisfaction, including how happy they are with their relationship, how frequently they disagree with their partner, and how they feel their relationship compares to others, using a 6- or 7-point Likert scale from 0 (e.g., Not at all true) to 5 or 6 (e.g., completely true). A total sum score is computed (range = 0 to 21) where higher scores indicate greater relationship satisfaction. The 4-item version has good psychometric properties and a cut-off for high relationship distress (Funk & Rogge, 2007).
Relationship Conflict | Baseline, 32-weeks gestation, and 4-, 8-, and 12-month follow-ups
  Relationship conflict will be measured using 2 items assessing conflict in the relationship from the Revised Dyadic Adjustment Scale (Busby, 1995). These items ask participants to report how often they argue with their partner or how often they get on each others' nerves. To measure sexual conflict, the same two items were adapted to ask specifically about sex. Participants respond using a Likert scale from 0 ("All the time) to 5 ("Never"). A total sum score is computed for each of relationship and sexual conflict (range = 0 to 10) where higher scores indicate less conflict.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: Yes
When publishing findings in scientific journals, the investigators will upload limited de-identified datasets specific to the analyses in question via the Open Science Framework (OSF) platform.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol will be published in a scientific journal while data collection is still ongoing. The datasets for each publication will be uploaded to OSF after the respective analysis is complete and will remain on OSF indefinitely.
Access Criteria: Researchers outside the research teams at Dalhousie University or the University of British Columbia will be able to access the uploaded datasets on the OSF. The data that will be shared on the OSF website will only contain the variables relevant to the analysis in question and will not contain any information that could identify the participants. Further, it will be password protected such that interested researchers will have to contact the research team for the password. Datasets may be inspected and analyzed by other researchers for the purposes of reproduction and verification of our findings, necessitating all responses included in the analysis to be included in the uploaded dataset.